CLINICAL TRIAL: NCT03612245
Title: Hygiene and Bucco-dental Status of Patients With Oral Streptococcal Endocarditis
Acronym: EI-DENTS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Bichat Hospital (Other); Central Hospital, Nancy, France (Other); CHU de Reims (Other); Pitié-Salpêtrière Hospital (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HC/2010/26
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective endocarditis (IE) is a rare (30 cases / million / year in France) and serious disease (20 % of deaths during hospitalization and 40 % after 5 years). The development of an IE results from the meeting between a bacteremia and a pre-existent heart disorder, most of the time valvular, allowing the transplant of the circulating bacteria and their multiplication in the endocardium. Recommendations of prophylactic antibiotic treatment have been established since 1954 for some medical, particularly dental procedures, at the origin of bacteremia. But this policy has recently been questioned because its efficacy has not been demonstrated.

The purpose of this study is identify the situations with risk, by comparing the oral health status and the hygiene of patients having an IE with oral streptococci to those in patients having an IE with microorganisms not of oral origin.

DETAILED DESCRIPTION:
It is a case-control observational study. The IE cases are recruited in hospitals participating to the french prospective observational "EI2008" cohort.

Cases are IE with oral streptococci whereas controls are IE with microorganisms not of oral origin.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Definite IE caused by oral streptococci (case) or by non-oral pathogens (control)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite IE treated in one of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
Oral health status | During the IE event
  Dental and periodontal evaluation by a dental surgeon or a stomatologist, according to a protocol of standardized examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duval X, Millot S, Chirouze C, Selton-Suty C, Moby V, Tattevin P, Strady C, Euvrard E, Agrinier N, Thomas D, Hoen B, Alla F; EI-dents Association pour l'Etude et la Prevention de l'Endocardite Infectieuse (AEPEI) Study Group. Oral Streptococcal Endocarditis, Oral Hygiene Habits, and Recent Dental Procedures: A Case-Control Study. Clin Infect Dis. 2017 Jun 15;64(12):1678-1685. doi: 10.1093/cid/cix237. PMID 28369398